CLINICAL TRIAL: NCT07047664
Title: Kidney Disease Sweat Sensor Patch for Early Diagnosis and Remote MonIToring
Brief Title: KERMIT: Sweat Patch for Early Kidney Disease Detection
Acronym: KERMIT
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Ioannina (Other)
Responsible Party: Principal Investigator, Evangelia Ntounousi, Ass. Prof. of Nephrology, Head of Nephrology Department, University of Ioannina
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: KERMIT-UOI-01; Horizon Europe EIC programme (Other Grant/Funding Number: Horizon Europe EIC programme)
Record Dates: First submitted 2025-06-03; First posted 2025-07-02 (Actual); Last update posted 2025-07-02 (Actual); Status verified 2025-06

CONDITIONS: Chronic Kidney Disease (CKD)
Keywords: CKD
MeSH Terms: conditions — Renal Insufficiency, Chronic

STUDY DESIGN:
Intervention Model Description: This is a non-randomized, parallel assignment interventional study designed to evaluate the diagnostic performance and safety of an experimental wearable sweat-sensing device. The study includes two parallel arms based on kidney function:
  * one arm of patients with chronic kidney disease (CKD) defined by an estimated glomerular filtration rate (eGFR) < 60 mL/min/1.73 m², and
  * one arm of patients with preserved eGFR (≥ 60 mL/min/1.73 m²) but with documented structural or functional kidney damage.
  All participants will undergo a single application of the wearable device, which non-invasively collects sweat to quantify kidney biomarkers.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- CKD with eGFR < 60 mL/min/1.73 m² (Other): CKD patients with reduced kidney function (eGFR < 60 mL/min/1.73 m²), and
  Interventions: Device: KERMIT dermal patch
- CKD with eGFR ≥ 60 mL/min/1.73 m²) (Other): CKD patients with preserved kidney function (eGFR ≥ 60 mL/min/1.73 m²) but with documented evidence of kidney damage (e.g., albuminuria, structural or genetic abnormalities).
  Interventions: Device: KERMIT dermal patch

INTERVENTIONS:
Device: KERMIT dermal patch — The KERMIT patch is a non-invasive, wearable device designed to collect sweat and measure concentrations of kidney function biomarkers, including creatinine, urea, and cystatin C. The patch integrates printed biosensors and a microfluidic system for electrochemical detection. It is applied to the skin for a short duration (typically <1 hour), with pilocarpine stimulation. This study evaluates the patch's performance in differentiating between CKD patients with reduced versus preserved renal function.
  Arms: CKD with eGFR < 60 mL/min/1.73 m²
Device: KERMIT dermal patch — The KERMIT patch is a non-invasive, wearable device designed to collect sweat and measure concentrations of kidney function biomarkers, including creatinine, urea, and cystatin C. The patch integrates printed biosensors and a microfluidic system for electrochemical detection. It is applied to the skin for a short duration (typically <1 hour), with pilocarpine stimulation. This study evaluates the patch's performance in differentiating between CKD patients with reduced versus preserved renal function.
  Arms: CKD with eGFR ≥ 60 mL/min/1.73 m²)

SUMMARY:
Chronic kidney disease (CKD) affects over 10% of the global population, leading to significant morbidity, mortality, and economic burden. Early detection is crucial for preventing disease progression and complications; however, awareness and diagnosis of CKD remain alarmingly low. Current methods rely on blood or urine analysis, which are invasive and require specialized facilities. The KERMIT patch aims to address this gap by providing a wearable lab-on-a-chip device capable of measuring key biomarkers from sweat non-invasively. This innovation has the potential to revolutionize CKD diagnosis, particularly in remote or underserved areas.

The KERMIT patch integrates functional printed biosensors, a high-frequency electrochemical microchip, and a sustainable microfluidic system. Sensors are fabricated using carbon inks and 2D materials, enabling immunodetection and non-enzymatic sensing of creatinine, urea, and cystatin C. Preliminary tests evaluated detection limits, skin compatibility, and carbon footprint.

ELIGIBILITY:
Inclusion Criteria:

Adults aged ≥18 years with stable CKD, defined as:

* eGFR < 60 mL/min/1.73 m², or
* eGFR ≥ 60 mL/min/1.73 m² with documented evidence of kidney damage (persistent albuminuria, structural abnormalities on imaging or histology, or genetic kidney disease).

Exclusion Criteria:

* Any signs of dermal infections, open wounds, or skin irritation.
* Significant variations in eGFR in the last two months, defined as any absolute change (either increase or decline) in eGFR of >10 mL/min/1.73m2 ;
* Patients with a functioning kidney graft;
* Patients receiving immunosuppression treatment;
* Patients with kidney stones;
* Patients with uncontrolled hypertension (a systolic blood pressure (SBP) >150 mmHg and/or diastolic blood pressure (DBP) >90 mmHg with measurements taken under standardized conditions (e.g after a 5-minute seated rest, using validated equipment);
* Patients receiving drugs reported to affect serum levels of creatinine and cystatin-c without affecting kidney function (i.e. cimetidine, trimethoprim, and fibrates);
* Known allergy to pilocarpine,
* Glaucoma;
* Patients with metal implants;
* Pregnancy;
* Active malignancy;
* Low life expectancy (<6 months) according to investigators judgement

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 52 (Estimated)
Dates: Start 2025-07-01 (Estimated); Primary Completion 2025-12 (Estimated); Study Completion 2026-07 (Estimated)

PRIMARY OUTCOMES:
Creatinine concentration in sweat | Day 1 (includes screening, device application, and sample analysis)
  Estimate the concentration of creatinine in sweat and assess its diagnostic accuracy in differentiating CKD patients with reduced kidney function (eGFR < 60 mL/min/1.73 m²) from those with preserved kidney function (eGFR ≥ 60 mL/min/1.73 m² but with documented kidney damage).
  Unit of Measure: µmol/L
Urea concentration in sweat | Day 1 (includes screening, device application, and sample analysis)
  Estimate the concentration of urea in sweat and assess its diagnostic accuracy in differentiating CKD patients with reduced kidney function (eGFR < 60 mL/min/1.73 m²) from those with preserved kidney function (eGFR ≥ 60 mL/min/1.73 m² but with documented kidney damage).
  Unit of Measure: mmol/L
Incidence of adverse events related to the wearable device | Day 1 (up to 1 hour post-device removal)
  Assess the number and severity of adverse events related to the use of the wearable sweat-sensing device, including skin irritation, discomfort, or allergic reactions.
  Unit of Measure: Number of events, graded by severity (mild, moderate, severe)